CLINICAL TRIAL: NCT04354051
Title: The Vascular Effects of Nitrite on Coronary Flow Under Normoxia and Hypoxia
Brief Title: The Nitrite and Coronary Flow Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of East Anglia (Other)
Collaborators: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 228798
Record Dates: First submitted 2020-02-10; First posted 2020-04-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Cardiovascular Diseases; Vasodilation; Hypoxia
MeSH Terms: conditions — Cardiovascular Diseases; Aneurysm; Hypoxia | interventions — Sodium Nitrite

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sodium nitrite (Experimental)
  Interventions: Drug: Sodium Nitrite

INTERVENTIONS:
Drug: Sodium Nitrite — Intravenous nitrite sodium infusion, dose 70μmol, of 5 minute duration (14μmol /min-1).

SUMMARY:
This study is a pharmacodynamic proof of concept study investigating the physiological effects of systemic infusion of nitrite on coronary blood flow using MRI.

DETAILED DESCRIPTION:
This is a healthy volunteer, proof of concept study.

The participant will have blood taken and this will be analysed for baseline levels of nitrate, nitrite and nitroso species. They will then have a baseline MRI to assess coronary flow in normoxia. Next, hypoxia will be induced using 12% oxygen/88% nitrogen. The participant will then have a baseline MRI to assess coronary flow in hypoxia (3 breath-hold image captures).

After all baseline images have been captured, the investigators will commence an intravenous nitrite sodium infusion, dose 70μmol, of 5 minute duration (14μmol /min-1). At the 5th minute, the participant have a further MRI image to assess coronary flow with the intervention in normoxia (3 breath-hold image captures).

A 10-minute washout will follow (with the half-life of nitrite being documented as 110 seconds). There will be optional repeat 3 breath-hold image captures at 5 minutes and at 10 minutes.

Next hypoxia will be induced using 12% oxygen/88% nitrogen again. The investigators will commence a second intravenous nitrite sodium infusion, dose 70μmol, 5 minute duration (14μmol /min-1). At the 5th minute, the participant will have a further MRI image to assess coronary flow with the intervention in hypoxia (3 breath-hold image captures).

At the end of the study the participant will have blood taken and this will be analysed for repeat levels of nitrate, nitrite and nitroso species.

All interventions will be performed by fully trained and competent medical staff.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged greater than or equal to 18 years
2. Not known to have any significant past medical history and not having regular follow up
3. Able to provide informed consent

Exclusion Criteria:

1. Significant medical, surgical or psychiatric disease that in the opinion of the Clinical Research Fellow would affect subject safety or significantly impact his/her ability to comply with follow-up. This would include any known clotting disorders.
2. Known allergy or intolerance to Nitrites
3. Known glucose-6-phosphate dehydrogenase (G6PD) deficiency or G6PD deficiency detected at screening in males of African, Asian or Mediterranean decent
4. Female subjects must be of non-childbearing potential, defined as follows: postmenopausal females who have had at least 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhoea with serum FSH>40mIU/ml or females who have had a hysterectomy, bilateral salpingectomy or bilateral oophorectomy at least 6 weeks prior to enrolment
5. Receipt of an investigational drug or biological agent within the 4 weeks prior to study entry or 5 times the drug half-life, whichever is the longer
6. Predisposed to acute on chronic limb ischemia evident from a history of claudication or known peripheral arterial disease
7. Any contra-indication to MRI, including the presence of an implanted metal device or suspected metal foreign bodies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
The effect of systemic sodium nitrite on the degree of vasorelaxation (captured by taking 4 sets of MRI images on the same study day, within a 2-hour window) in the coronary vessels in normoxia and hypoxia in healthy participants | All data and images collected on study day within a 2-hour time window. All study days are now complete.
  This will be measured on the study day through the acquisition of 4 set of separate MRI images (each image set acquisition duration 3-5 minutes). 4 conditions for image acquisition: normoxia without nitrite, hypoxia without nitrite, normoxia with nitrite and hypoxia with nitrite. Images captured using coronary MRI.

SECONDARY OUTCOMES:
The change in systemic levels of nitrate, nitrite and nitroso species after intravenous sodium nitrite infusion | Anticipated within 1 year of study completion
  This is anticipated to take place within 1 year of completion of the study via ozone-based chemiluminescence or high performance liquid chromatography. The data will show the change in nitrate, nitrite and nitroso species levels in the study participants plasma before and after the nitrite infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Frenneaux, FRCP (UK), Principal Investigator — University of East Anglia
Locations (1):
- University of East Anglia, Norwich, Norfolk, United Kingdom

IPD SHARING:
Plan to Share IPD: No